CLINICAL TRIAL: NCT02779881
Title: Epigenetic Features of FoxP3 in Children With Cow's Milk Allergy
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Federico II University
Other Study IDs: 1-14
Record Dates: First submitted 2016-05-16; First posted 2016-05-23 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Cow's Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Healthy controls: Healthy controls
- Children at diagnosis of cow's milk allergy: Children at diagnosis of cow's milk allergy
- Subjects outgrown cow's milk allergy with formula+probiotic: Tolerant with extensively hydrolyzed casein formula with Lactobacillus rhamnosus GG
  Interventions: Dietary Supplement: Extensively hydrolyzed casein formula plus LGG
- Subjects outgrown cow's milk allergy assuming other formulas: Subjects tolerant with other formulas

INTERVENTIONS:
Dietary Supplement: Extensively hydrolyzed casein formula plus LGG
  Groups: Subjects outgrown cow's milk allergy with formula+probiotic

SUMMARY:
Epigenetic mechanisms have been implicated in the pathogenesis of food allergy. The investigators previously demonstrated that tolerance acquisition in children with Immunoglobulin E- (IgE) mediated cow's milk allergy (CMA) is driven by epigenetic modulation of the Th1 and Th2 cytokine genes. A regulatory T cell (Treg) suppressive phenotype, characterized by stable expression of the transcription factor "Forkhead box Protein 3" (FoxP3), plays a pivotal role in food tolerance. FoxP3 mRNA expression is lower in children with atopic asthma or IgE-mediated food allergy than in healthy children. FoxP3 stable expression requires full CpG demethylation of its transcriptional regulatory regions, and, moreover, hypermethylation of the FoxP3 gene has been associated with reduced Treg function and allergy.

DNA methylation is a biologically and chemically stable epigenetic modification that locks in long-term gene expression patterns. The demethylation status of FoxP3 at a highly conserved region within the Treg-specific-demethylated-region (TSDR), a CpG-rich, located on the 2nd conserved non-coding sequence of FoxP3 (CNS2), is restricted to Tregs. Transcriptional activity of the TSDR is essentially determined by its methylation status : it is completely inactive in its methylated state, but when the TSDR is demethylated, transcription factors such as Ets-1 and Creb can bind to the TSDR. TSDR demethylated and open chromatin conformation in the Foxp3 locus leads to stable phenotype differentiated Foxp3+ Treg. FoxP3 TSDR demethylation in peripheral blood mononuclear cells (PBMCs) has been associated with reduced atopic sensitization and asthma in children. Epigenetic regulation of antigen-induced T-cell subsets may predict a state of immune tolerance in food allergy. Indeed, DNA methylation of the FoxP3 gene in Tregs decreased during oral tolerance acquisition in patients with peanut allergy undergoing oral immunotherapy. The aim of this study was to evaluate further the epigenetic regulation of FoxP3 gene in children with IgE-mediated CMA.

ELIGIBILITY:
Inclusion Criteria:

* IgE-mediated CMA children (aged 3 to 18 months)

Exclusion Criteria:

* allergic disorders or food allergies other than cow's milk allergy
* eosinophilic disorders of the gastrointestinal tract
* food protein-induced enterocolitis syndrome
* concomitant chronic systemic diseases
* congenital cardiac defects
* active tuberculosis
* autoimmune diseases
* immunodeficiency
* chronic inflammatory bowel diseases
* celiac disease
* cystic fibrosis
* metabolic diseases
* lactose intolerance
* malignancy
* chronic pulmonary diseases
* malformations of the gastrointestinal tract

Ages: 3 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: IgE-mediated CMA children (aged 3 to 18 months) consecutively referred to the tertiary Pediatric Allergy Center for oral food challenge.
  During the same study period, consecutive healthy children, not at risk of atopic disorders (namely, those without a first-degree relative affected by an atopic disorder), attending the Center because of minimal surgical procedures served as a control group.
  A venous blood sample (4 ml) was obtained from all patients after oral challenge.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
DNA demethylation (rate, in %) of the Treg-specific-demethylated-region (TSDR) of FoxP3 | At enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paparo L, Nocerino R, Cosenza L, Aitoro R, D'Argenio V, Del Monaco V, Di Scala C, Amoroso A, Di Costanzo M, Salvatore F, Berni Canani R. Epigenetic features of FoxP3 in children with cow's milk allergy. Clin Epigenetics. 2016 Aug 12;8:86. doi: 10.1186/s13148-016-0252-z. eCollection 2016. PMID 27525046